CLINICAL TRIAL: NCT01191229
Title: Prospective Evaluation of Visual Outcomes With Tecnis One-Piece Multifocal Intraocular Lenses Compared With Patients Previously Implanted With Crystalens AO
Brief Title: Prospective Evaluation of Visual Outcomes With Tecnis One-Piece Multifocal Intraocular Lenses Compared With Patients Previously Implanted With Crystalens Aspheric Optic (AO)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Mitch Jackson, MD, JacksonEye
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tecnis One-Piece MF IOL
Record Dates: First submitted 2010-08-19; First posted 2010-08-30 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: To Collect Information About Visual Outcomes and Participant Satisfaction

ARMS (2):
- Tecnis One-Piece MF IOL (No Intervention): It is planned that about 25 people who are at least 18 years old who are scheduled to have the Tecnis One-Piece Multifocal Intraocular Lenses placed into their eyes after cataract surgery
  Interventions: Device: Tecnis one-piece MF IOL
- Crystalens AO (No Intervention): It is planned that about 25 people who are at least 18 years old and have been implanted with Crystalens AO
  Interventions: Device: Crystalens AO

INTERVENTIONS:
Device: Tecnis one-piece MF IOL — 25 patients to be implanted after cataract surgery
  Arms: Tecnis One-Piece MF IOL
Device: Crystalens AO — 25 patients that are previously implanted
  Arms: Crystalens AO

SUMMARY:
The study is being conducted to collect information about visual outcomes and participant satisfaction with the Tecnis One-Piece Multifocal (MF) Intraocular Lenses (IOLs) compared with participants previously implanted with Crystalens Aspheric Optic (AO) IOLs. The U.S. Food and Drug Administration (FDA) has cleared the Tecnis One-Piece MF IOL for visual correction of aphakia (replacing a removed lens in the eye) in adults.

ELIGIBILITY:
Inclusion Criteria:

* Key Inclusion Criteria for Part 1:

  * Age 18 or greater
  * Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation has been planned for both eyes
  * Visual potential of 20/30 or better in each eye after cataract removal and IOL implantation
  * Preoperative best-corrected distance visual acuity (BCDVA) worse than 20/40 Snellen
  * Naturally dilated pupil size (in dim light) > 3.5 mm (with no dilation medications) for both eyes
  * Preoperative corneal astigmatism of 1.5 D or less
  * Clear intraocular media other than cataract
  * Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Inclusion Criteria for Part 2

* At least 18 years of age
* Underwent bilateral implantation with Crystalens AO at least 6 months previously
* Visual potential of 20/30 or better in each eye after cataract removal and IOL implantation
* Preoperative best-corrected distance visual acuity (BCDVA) worse than 20/40 Snellen
* Naturally dilated pupil size (in dim light) > 3.5 mm (with no dilation medications) for both eyes
* Preoperative corneal astigmatism of 1.5 D or less
* Clear intraocular media other than cataract
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Key Exclusion Criteria for Part 1:

  * Use of systemic or ocular medications that may affect vision
  * Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus, immunocompromised, etc.)
  * Subjects with diabetes mellitus
  * Uncontrolled systemic or ocular disease
  * History of ocular trauma or prior ocular surgery
  * Amblyopia or strabismus
  * Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
  * Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
  * Patients with forme fruste keratoconus or keratoconus
  * Subjects who may be expected to require retinal laser treatment or other surgical intervention
  * Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
  * Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 4.0 mm under mesopic/scotopic conditions)
  * Contact lens usage within 6 months for PMMA contacts lenses, 1 month for gas permeable lenses or 1 week for extended-wear and daily-wear soft contact lenses
  * Requiring an intraocular lens <15.0 or >26.0 diopters

Exclusion Criteria for Part 2

* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
* Patients with forme fruste keratoconus or keratoconus
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 4.0 mm under mesopic/scotopic conditions)
* Requiring an intraocular lens <15.0 or >26.0 diopters Exclusion Criteria for Part 2
* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
* Patients with forme fruste keratoconus or keratoconus
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 4.0 mm under mesopic/scotopic conditions)
* Requiring an intraocular lens <15.0 or >26.0 diopters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incision size | 1 year
  Part 1 Only:
  The primary outcome measure is incision size at three points:
  Immediately after application of the keratome blade Post phacoemulsification Post Tecnis IOL implantation Target refraction vs. achieved
  Part 1 and 2:
  UCVA data at distance, intermediate, and near Near vision will be measured in mesopic and photopic conditions standardized with light meter BCVA at distance and near Enhancement rates Spectacle independence questionnaire and patient satisfaction Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- JacksonEye, Lake Villa, Illinois, United States